CLINICAL TRIAL: NCT02707016
Title: Emergence Delirium in Children: a Randomized Clinical Trial of Different Doses of Sevoflurane During Induction of Anesthesia
Brief Title: Different Doses of Sevoflurane During Induction of Anesthesia on Emergence Delirium in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15-153
Record Dates: First submitted 2016-03-07; First posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Delirium
Keywords: Emergence delirium; Sevoflurane; Pediatric anesthesia
MeSH Terms: conditions — Delirium; Emergence Delirium | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose sevoflurane (Other): Inhaled sevoflurane 8% during induction of general anesthesia (from the start of gas administration to the insertion of a laryngeal mask).
  After laryngeal mask insertion, sevoflurane will be reduced to 4%. Caudal block with L-bupivacaine 0.25% will be performed in all children.
  After caudal block, sevoflurane will be reduced to 0.75 MAC according to age of the child and maintained until the end of surgery After surgery, PAED and pain scales will be administered every 15 minutes up to 2 hours after surgery.
  Interventions: Other: Sevoflurane 8%
- Low dose sevoflurane (Other): Inhaled sevoflurane 5% during induction of general anesthesia (from the start of gas administration to the insertion of a laryngeal mask).
  After laryngeal mask insertion, sevoflurane will be reduced to 4%. Caudal block with L-bupivacaine 0.25% will be performed in all children.
  After caudal block, sevoflurane will be reduced to 0.75 MAC according to age of the child and maintained until the end of surgery After surgery, PAED and pain scales will be administered every 15 minutes up to 2 hours after surgery.
  Interventions: Other: Sevoflurane 5%

INTERVENTIONS:
Other: Sevoflurane 8% — Sevoflurane 8% (high dose) during anesthesia induction
  Other Names: Sevorane
  Arms: High dose sevoflurane
Other: Sevoflurane 5% — Sevoflurane 5% (low dose) during anesthesia induction
  Other Names: Sevorane
  Arms: Low dose sevoflurane

SUMMARY:
The investigators aim to reduce the incidence of emergence delirium in children aged 2-7 years old by using two different doses of sevoflurane during inhalatory induction of anesthesia.

DETAILED DESCRIPTION:
Sevoflurane is an inhalational agent widely used in general anesthesia, both for induction and maintenance of anesthesia. It is not irritative on the airways and has a pleasant smell. Within their properties are: low partition coefficient blood / gas (rapid induction and awakening), low heart, liver and kidney toxicity. Inhalational induction in pediatric anesthesia with this agent is frequent to avoid vein puncture in awake patients and is generally done with maximum doses available to obtain a fast loss of consciousness.

Emergence delirium (ED) is frequent in children. It is defined as a mental disorder during recovery from general anesthesia that may include hallucinations, delusions and confusion expressed by crying, restlessness and involuntary physical activity. It usually lasts for 30 minutes and is not necessarily related to pain. During this episodes, children can hurt themselves or others, lose vascular catheters or other invasive devices. ED can generate anxiety and stress in caretakers, delay transfer from Post-Anesthesia Care Units (PACU), increase costs of medical attention and increase use of opioids or other sedatives.

Many interventions have been used to decrease the appearance of ED such as dexmedetomidine, clonidine, benzodiazepines, propofol among others but with no consistent results. The use of sevoflurane has been linked with ED in children and it can induce seizures in high doses (over 2 MAC).

The aim of this study is to test whether using a lower dose of sevoflurane (5%) during induction of anesthesia in children results in less ED than using higher doses (8%).

ELIGIBILITY:
Inclusion Criteria:

* Surgery with caudal block: circumcision (phimosis), hernioplasty (inguinal hernia)
* American Society of Anesthesiologists (ASA) classification of I or II

Exclusion Criteria:

* Use of Total Intravenous Anesthesia (TIVA)
* Familiar or personal history of Malignant Hyperthermia
* Contraindication to caudal block
* Parents or legal guardians do not sign informed consent

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Emergence delirium | From end of gas administration up to 2 hours after surgery
  Emergence delirium will be evaluated with the Pediatric Anesthesia Emergence Delirium scale every 15 minutes

SECONDARY OUTCOMES:
Pain | From end of gas administration up to 2 hours after surgery
  Pain will be evaluated according to age of children: CHIPPS scale for under 3 years, faces for children between 4 and 6 years old, Visual Analogue Scale (VAS) with older children.
Bispectral Index | From start of induction until end of surgery
  Bispectral Index (BIS) monitoring will be used during surgery and recorded at following times: after insertion of IV access, after insertion of laryngeal mask, after caudal block, after lowering dose of sevoflurane to 0.75 MAC, after skin incision, at the end of surgery
Heart rate | From start of induction until end of surgery
  Measured with pulse oximetry, recorded at following times: after insertion of IV access, after insertion of laryngeal mask, after caudal block, after lowering dose of sevoflurane to 0.75 MAC, after skin incision, at the end of surgery
Blood pressure | From start of induction until end of surgery
  Measured with non-invasive blood pressure cuff, recorded at following times: after insertion of IV access, after insertion of laryngeal mask, after caudal block, after lowering dose of sevoflurane to 0.75 MAC, after skin incision, at the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Aeschlimann, MD, Principal Investigator — Assistant Professor
Locations (1):
- División de Anestesia - Facultad de Medicina Pontificia Universidad Católica, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bajwa SA, Costi D, Cyna AM. A comparison of emergence delirium scales following general anesthesia in children. Paediatr Anaesth. 2010 Aug;20(8):704-11. doi: 10.1111/j.1460-9592.2010.03328.x. PMID 20497353
- [Background] Li X, Xia Q, Li W. Comparison of the effects of dezocine, fentanyl, and placebo on emergence agitation after sevoflurane anesthesia in children. Int J Clin Pharmacol Ther. 2015 Mar;53(3):241-6. doi: 10.5414/CP202184. PMID 25669611
- [Background] Oofuvong M, Siripruekpong S, Naklongdee J, Hnookong R, Lakateb C. Comparison the incidence of emergence agitation between sevoflurane and desflurane after pediatric ambulatory urologic surgery. J Med Assoc Thai. 2013 Nov;96(11):1470-5. PMID 24428097
- [Background] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Background] Ozcan A, Kaya AG, Ozcan N, Karaaslan GM, Er E, Baltaci B, Basar H. [Effects of ketamine and midazolam on emergence agitation after sevoflurane anaesthesia in children receiving caudal block: a randomized trial]. Rev Bras Anestesiol. 2014 Nov-Dec;64(6):377-81. doi: 10.1016/j.bjan.2014.01.004. Epub 2014 Aug 29. Portuguese. PMID 25437692
- [Background] Saxena A, Sethi A, Agarwal V, Godwin RB. Effect of caudal clonidine on emergence agitation and postoperative analgesia after sevoflurane anaesthesia in children: Randomised comparison of two doses. Indian J Anaesth. 2014 Nov-Dec;58(6):719-25. doi: 10.4103/0019-5049.147163. PMID 25624536
- [Background] Abdel-Ma'boud MA. Effect of dexemeditomedine and propofol on the prevention of emergence agitation following sevoflurane anesthesia in Egyptian children. J Egypt Soc Parasitol. 2014 Dec;44(3):687-94. doi: 10.12816/0007872. PMID 25643510
- [Background] Zhang C, Hu J, Liu X, Yan J. Effects of intravenous dexmedetomidine on emergence agitation in children under sevoflurane anesthesia: a meta-analysis of randomized controlled trials. PLoS One. 2014 Jun 16;9(6):e99718. doi: 10.1371/journal.pone.0099718. eCollection 2014. PMID 24932765
- [Background] Costi D, Cyna AM, Ahmed S, Stephens K, Strickland P, Ellwood J, Larsson JN, Chooi C, Burgoyne LL, Middleton P. Effects of sevoflurane versus other general anaesthesia on emergence agitation in children. Cochrane Database Syst Rev. 2014 Sep 12;2014(9):CD007084. doi: 10.1002/14651858.CD007084.pub2. PMID 25212274
- [Background] Dahmani S, Delivet H, Hilly J. Emergence delirium in children: an update. Curr Opin Anaesthesiol. 2014 Jun;27(3):309-15. doi: 10.1097/ACO.0000000000000076. PMID 24784918
- [Background] Gibert S, Sabourdin N, Louvet N, Moutard ML, Piat V, Guye ML, Rigouzzo A, Constant I. Epileptogenic effect of sevoflurane: determination of the minimal alveolar concentration of sevoflurane associated with major epileptoid signs in children. Anesthesiology. 2012 Dec;117(6):1253-61. doi: 10.1097/ALN.0b013e318273e272. PMID 23103557
- [Background] Schultz B, Otto C, Schultz A, Osthaus WA, Krauss T, Dieck T, Sander B, Rahe-Meyer N, Raymondos K. Incidence of epileptiform EEG activity in children during mask induction of anaesthesia with brief administration of 8% sevoflurane. PLoS One. 2012;7(7):e40903. doi: 10.1371/journal.pone.0040903. Epub 2012 Jul 19. PMID 22829896
- [Background] Kreuzer I, Osthaus WA, Schultz A, Schultz B. Influence of the sevoflurane concentration on the occurrence of epileptiform EEG patterns. PLoS One. 2014 Feb 26;9(2):e89191. doi: 10.1371/journal.pone.0089191. eCollection 2014. PMID 24586585
- [Background] Pilge S, Jordan D, Kochs EF, Schneider G. Sevoflurane-induced epileptiform electroencephalographic activity and generalized tonic-clonic seizures in a volunteer study. Anesthesiology. 2013 Aug;119(2):447. doi: 10.1097/ALN.0b013e31827335b9. No abstract available. PMID 23221897
- [Background] Julliac B, Cotillon P, Guehl D, Richez B, Sztark F. Target-controlled induction with 2.5% sevoflurane does not avoid the risk of electroencephalographic abnormalities. Ann Fr Anesth Reanim. 2013 Oct;32(10):e143-8. doi: 10.1016/j.annfar.2013.07.812. Epub 2013 Sep 12. PMID 24035611
- [Background] Hadi SM, Saleh AJ, Tang YZ, Daoud A, Mei X, Ouyang W. The effect of KETODEX on the incidence and severity of emergence agitation in children undergoing adenotonsillectomy using sevoflurane based-anesthesia. Int J Pediatr Otorhinolaryngol. 2015 May;79(5):671-6. doi: 10.1016/j.ijporl.2015.02.012. Epub 2015 Feb 19. PMID 25770644
- [Background] Adachi M, Ikemoto Y, Kubo K, Takuma C. Seizure-like movements during induction of anaesthesia with sevoflurane. Br J Anaesth. 1992 Feb;68(2):214-5. doi: 10.1093/bja/68.2.214. PMID 1540467
- [Background] Vakkuri A, Yli-Hankala A, Sarkela M, Lindgren L, Mennander S, Korttila K, Saarnivaara L, Jantti V. Sevoflurane mask induction of anaesthesia is associated with epileptiform EEG in children. Acta Anaesthesiol Scand. 2001 Aug;45(7):805-11. doi: 10.1034/j.1399-6576.2001.045007805.x. PMID 11472278
- [Background] Yli-Hankala A, Vakkuri A, Sarkela M, Lindgren L, Korttila K, Jantti V. Epileptiform electroencephalogram during mask induction of anesthesia with sevoflurane. Anesthesiology. 1999 Dec;91(6):1596-603. doi: 10.1097/00000542-199912000-00009. PMID 10598599
- [Background] Vakkuri A, Jantti V, Sarkela M, Lindgren L, Korttila K, Yli-Hankala A. Epileptiform EEG during sevoflurane mask induction: effect of delaying the onset of hyperventilation. Acta Anaesthesiol Scand. 2000 Jul;44(6):713-9. doi: 10.1034/j.1399-6576.2000.440609.x. PMID 10903015
- [Background] Voepel-Lewis T, Malviya S, Tait AR. A prospective cohort study of emergence agitation in the pediatric postanesthesia care unit. Anesth Analg. 2003 Jun;96(6):1625-1630. doi: 10.1213/01.ANE.0000062522.21048.61. PMID 12760985
- [Background] Aouad MT, Kanazi GE, Siddik-Sayyid SM, Gerges FJ, Rizk LB, Baraka AS. Preoperative caudal block prevents emergence agitation in children following sevoflurane anesthesia. Acta Anaesthesiol Scand. 2005 Mar;49(3):300-4. doi: 10.1111/j.1399-6576.2005.00642.x. PMID 15752392
- [Background] Welborn LG, Hannallah RS, Norden JM, Ruttimann UE, Callan CM. Comparison of emergence and recovery characteristics of sevoflurane, desflurane, and halothane in pediatric ambulatory patients. Anesth Analg. 1996 Nov;83(5):917-20. doi: 10.1097/00000539-199611000-00005. PMID 8895263